CLINICAL TRIAL: NCT06498609
Title: Assessment of the Efficacy of Microosteoperforations Versus Injectable Platelet-rich Fibrin During Orthodontic Leveling and Alignment of Mandibular Incisors: A Comparative Clinical Trial
Brief Title: Assessment of the Efficacy of Microosteoperforations Versus Injectable Platelet-rich Fibrin During Orthodontic Leveling and Alignment of Mandibular Incisors
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, principal investigator, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1001/3560
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-05

CONDITIONS: Effect of Platelet Rich Fibrin Versus Microosteoperforation Compaed to Control Group Toothmovement
MeSH Terms: interventions — morpholinopropane sulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microosteoperforation (Experimental): MOPs with leveling and alignment that will be performed tow time according to standardized protocol
  Interventions: Procedure: MOPs with leveling and alignment
- Injectable platelet rich fibrin (Experimental): i-PRF with leveling and alignment that will be performed tow time according to standardized protocol
  Interventions: Biological: iprf
- control group (No Intervention): leveling and alignment that will be performed without any intervention

INTERVENTIONS:
Biological: iprf — i-PRF with leveling and alignment
  Arms: Injectable platelet rich fibrin
Procedure: MOPs with leveling and alignment — mop
  Arms: Microosteoperforation

SUMMARY:
The aim of this prospective clinical study will be to compare the efficacy of micro osteoperforations versus injectable platelet-rich fibrin during orthodontic leveling and alignment of mandibular incisors.

ELIGIBILITY:
Inclusion Criteria:

1. An age range from 15 to 25 years.
2. Participants who had a full set of permanent dentitions excluding the third molar.
3. Participants who had moderate crowding in the mandibular arch according to Little's irregularity index that necessitates non-extraction treatment in the mandibular arch.
4. Normal vertical facial proportions.
5. Participants who had good oral hygiene and no periodontal disease.
6. No systemic diseases or regular medication that could interfere and/or affect orthodontic teeth movement.
7. No evidence of craniofacial anomalies, such as clef lip and palate or previous history of trauma, bruxism, or parafunction.
8. No tooth size, shape, or root abnormalities visible on patient's radiographic records.

Exclusion Criteria:

1. Previous orthodontic treatment.
2. Any skeletal dysplasia or craniofacial malformation.
3. Retained primary or missing permanent teeth in the anterior area, and any kind of tooth/root shape anomaly or history of trauma affecting the incisors.
4. Systemic diseases or regular use of medications that could interfere with OTM.
5. Patients with root resorption, impacted canines, or dental anomalies.
6. Poor oral hygiene and uncontrolled periodontal diseases.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
assessment of acceleration of leveling and alignment of mandibular incisors | post interventional at 4months
  rate of leveling and alignment

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Fares, Student, Principal Investigator — Al-Azhar University
Locations (1):
- Alazhar University, Cairo, Egypt